CLINICAL TRIAL: NCT01492049
Title: Pilot Trial - Promoting Health Literacy for Colorectal Cancer Screening
Brief Title: R-21 Colorectal Cancer Screening (CRCS) Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2010-0698; R21CA132669 (NIH); NCI-2015-01899 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Promoting Health Literacy; Patient education program; Colorectal Cancer Screening; CRCS; Patient decision aid; PtDA; Video; Questionnaires; Surveys
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (PtDA) (Experimental): Participants view Patient decision aid (PtDA) video.
  Interventions: Behavioral: CRCS patient decision aid (PtDA) video; Behavioral: Questionnaires
- Control (Active Comparator): Participants view a video on Essential Hypertension.
  Interventions: Behavioral: Questionnaires; Behavioral: Essential Hypertension video

INTERVENTIONS:
Behavioral: CRCS patient decision aid (PtDA) video — Participant views PtDA program video in same room as research assistant who offers instruction as needed.
  Arms: Patient Decision Aid (PtDA)
Behavioral: Questionnaires — Up to 3 questionnaires (baseline demographics, post-intervention evaluation, and follow up) taking from 5 to 25 minutes to complete each.
  Other Names: survey
Behavioral: Essential Hypertension video — Participant views Essential Hypertension video in same room as research assistant who offers instruction as needed.
  Arms: Control

SUMMARY:
The goal of this study is to test patient education program for decision making about colorectal cancer (CRC) screening in community health centers.

DETAILED DESCRIPTION:
Baseline Visit:

If you agree to take part in this study, you will complete a questionnaire that asks demographic questions (such as your age and sex) and questions about colorectal cancer. It should take about 10-15 minutes to complete.

You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. If you are in Group 1, you will view a colorectal cancer program. If you are in Group 2, you watch a program on Essential Hypertension.

You will watch the program on a laptop in the clinic. The program is about 30 minutes long. After you watch the program, you will complete a questionnaire that asks what you thought about the program and some questions about understanding medical information. It should take about 5-10 minutes to complete the questionnaire.

You will be called 1-3 weeks after your baseline visit to complete a questionnaire by phone. The call should last about 20-25 minutes. You will be asked if you discussed colorectal cancer screening tests with your doctor, your preferences for colorectal cancer screening tests, and if any colorectal cancer screening tests were ordered.

At Month 3, your medical record will be reviewed by the study staff.

Length of Study:

You will be off study after your medical record is reviewed at Month 3.

This is an investigational study.

Up to 180 participants (90 Hispanic and 90 African-American) will take part in this study. All participants will be enrolled from the Harris County Hospital District and Kelsey-Seybold outpatient clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients
2. 49 -75 years of age
3. English-speaking African American or Spanish-speaking Hispanic patients (upon approval of spanish language arm)

Exclusion Criteria:

1. History of colorectal cancer
2. History of polyps
3. Any inflammatory bowel disease (IBD), e.g. Crohn's disease or ulcerative colitis
4. Family history of colorectal cancer in a first degree relative
5. Had fecal occult blood test (FOBT) in the past year, flexible sigmoidoscopy in the past 5 years or colonoscopy in the past 10 years

Ages: 49 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer screening (CRCS) Rate of Participants | 24 months for study duration
  CRCS rates in the patient decision aid and control subjects based on medical record reviews, physician orders for screening endoscopy after the baseline visit also from medical record reviews, and intentions to complete CRCS based on self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Harris County Hospital District, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org